CLINICAL TRIAL: NCT03559439
Title: CD19-targeting CAR T Cell Therapy in the Treatment of Relapsed or Refractory CD19 Positive B-cell Malignancies
Brief Title: CD19-targeting CAR T Cells in Relapsed or Refractory CD19 Positive B-cell Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Tong Ren Hospital (Other)
Collaborators: Gracell Biotechnology Ltd. (Other)
Responsible Party: Principal Investigator, Liu Ligen, Principal Investigator, Shanghai Tong Ren Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTA001
Record Dates: First submitted 2018-05-30; First posted 2018-06-18 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: B-cell Malignancy; B-cell Lymphoma; B-Cell Acute Lymphoblastic Leukaemia
MeSH Terms: conditions — Lymphoma, B-Cell; Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19 CAR T (Experimental): CD19 CAR T cells transduced with a lentiviral vector to express anti-CD19 scFv CD3z:CD28 administered by IV infusion.
  Interventions: Biological: CD19 CAR T

INTERVENTIONS:
Biological: CD19 CAR T — CD19 CAR T cells transduced with a lentiviral vector to express anti-CD19 scFv CD3z:CD28 administered by IV infusion. Subjects will receive 0.1-10 x 10^6 transduced CAR T cells as a split dose over three days as follows:Day 1, 10% fraction, Day 2, 30% fraction, Day 3, 60% fraction.

SUMMARY:
This is a single center, single arm, open-label phase 1 study to determine the safety and efficacy of autologous T cells expressing CD19 chimeric antigen receptors in adults with CD19+ B cell malignancies.

DETAILED DESCRIPTION:
This is a single-center, Open Label phase I clinical trial, 9 subjects planned to be enrolled. The subjects will be divided into low-dose group, medium-dose group and high-dose group.Dose CAR+ cells/kg Low 1×105 Medium 2×106 High 6×106

ELIGIBILITY:
Inclusion Criteria:

1. CD19+ relapsed or refractory B cell malignancies:

   * Relapsed or refractory B acute lymphocytic leukemia.

     * Relapse was defined as presence of > 5% blasts at screening, or second or subsequent bone marrow relapse, or any bone marrow relapse after allogeneic stem cell transplant and must be ≥ 6 months from stem cell transplant at the time of infusion.
     * Refractory was defined by not achieving an initial complete response after 2 cycles of a standard chemotherapy regimen . Patients who were refractory to subsequent chemotherapy regimens after an initial remission were considered chemorefractory
   * Patients with Ph+ acute lymphocytic leukemia were eligible if they are intolerant to or have not achieved a remission after two lines of tyrosine kinase inhibitor therapy, or if tyrosine kinase inhibitor therapy is contraindicated, or ineligible for allogeneic stem cell transplant because of:

     * Comorbid disease
     * Other contraindications to allogeneic stem cell transplant conditioning regimen
     * Lack of suitable donor
     * Prior hematopoietic stem cell transplant
     * Declined allogeneichematopoietic stem cell transplant as a therapeutic option
   * Relapsed or refractory non-Hodgkin's lymphoma

     * Histopathological CD19+.
     * No response to last line of therapy i. partial response as best response to most recent therapy regimen ii. partial response as best response to most recent therapy with duration no longer than 6 month from last dose of therapy
     * Refractory post-Autologous stem cell transplant i. Disease progression or relapsed less than or equal to 12 months of Autologous stem cell transplant (must have biopsy proven recurrence in relapsed subjects) ii. If salvage therapy is given post-Autologous stem cell transplant, the subject must have had no response to or relapsed after the last line of therapy
     * Subjects must have received adequate prior therapy including at a minimum: anti-CD20 monoclonal antibody unless investigator determines that tumor is CD20-negative and an anthracycline containing chemotherapy regimen for subjects with transformed follicular lymphoma must have received prior chemotherapy for follicular lymphoma and subsequently have chemorefractory disease after transformation to Diffuse large B-cell lymphoma
   * At least one measurable lesion per revised IWG Response Criteria
2. 18-75 years old
3. Expected survival ≥ 12 weeks
4. Adequate renal, hepatic, pulmonary and cardiac function defined as:

   * Creatinine clearance (as estimated by Cockcroft Gault) > 60 mL/min
   * Serum ALT/AST <2.5 ULN
   * Total bilirubin <1.5 mg/dl, except in subjects with Gilbert's syndrome
   * Cardiac ejection fraction >50%, no evidence of pericardial effusion as determined by an echocardiogram, and no clinically significant pleural effusion
   * Baseline oxygen saturation >92% on room air
5. Eastern cooperative oncology group (ECOG) performance status of 0 - 2
6. Pregnant or lactating women must have a negative pregnancy test before infusion, and agree to take effective contraception during the trial
7. Apheresis product received and accepted
8. Written informed consent

Exclusion Criteria:

1. Isolated extra-medullary relapse leukemia
2. Other malignancies
3. Concomitant genetic syndrome, with the exception of Down Syndrome
4. Burkitt's lymphoma/leukemia
5. Treatment with any prior gene therapy product, anti-CD19/anti-CD3 therapy, or any other anti-CD19 therapy
6. Active hepatitis B, C, or any uncontrolled infection
7. Grade 2 to 4 Graft versus Host Disease (GVHD)
8. Medications or treatments that were to be excluded:

   * Corticosteroids within 72 hours of infusion, with the exception of physiologic replacement
   * Allogeneic cellular therapy, such as donor lymphocyte infusion within 6 weeks prior to infusion
   * Graft versus Host Disease therapies
   * Chemotherapy stopped prior to lymphodepletion based on clearance
   * central nervous system prophylaxis treatment
9. Active central nervous system disease (central nervous system 2 disease [Cerebral spinal fluid containing blasts, but < 5 WBCs/microliter] patients were eligible)
10. Any condition that investigator considered may increase the risk of the subjects or interfere with the trial results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2018-04-24 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of toxicities and adverse events | 24 weeks
  To assess the frequency and severity of toxicities and adverse events according to NCI CTC v4.0

SECONDARY OUTCOMES:
overall response rate | 24 week
  To assess the overall response rate after CD19 CAR T infusion in R/R B cell malignancies
overall survival | 24 week
  To assess the overall survival in patients with R/R B cell malignancies

CONTACTS AND LOCATIONS:
Overall Officials: Ligen Liu, Principal Investigator — Shanghai Tong Ren Hospital
Locations (1):
- Shanghai Tong Ren hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No